CLINICAL TRIAL: NCT07035444
Title: Enteral Nutrition Supplemented With L-Carnitine for Cachexia in Non-Small Cell Lung Cancer: A Randomized Controlled Trial
Brief Title: Enteral Nutrition With L-Carnitine for Cachexia in Non-Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZXZYTSLC05
Record Dates: First submitted 2025-06-05; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-05

CONDITIONS: Non-Small Cell Lung Cancer; Cachexia
Keywords: L-carnitine; Enteral nutrition
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Cachexia | interventions — Carnitine; Enteral Nutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enteral nutrition (Active Comparator): During the entire study period (84 days), research participants will receive 500 ml of enteral nutrition solution daily. The nutrition is provided in two 55 g packets of nutritional powder. Each packet is dissolved in 220 ml of warm boiled water at 55°C to prepare 250 ml of the nutrition solution. Depending on the individual circumstances of the research participants, the solution can be taken in 2 to 3 divided doses daily, with a total daily volume of 500 ml.
  Interventions: Dietary Supplement: Enteral Nutrition
- Enteral Nutrition with L-Carnitine (Experimental): During the entire study period (84 days), research participants will receive 500 ml of enteral nutrition solution containing 4 g of L-carnitine daily. The nutrition consists of two 55 g packets of nutritional powder. Each packet is dissolved in 220 ml of warm boiled water at 55°C to make 250 ml of the nutrition solution. Depending on the individual situation of the research participants, the solution can be taken in two to three divided doses daily, with a total daily volume of 500 ml
  Interventions: Dietary Supplement: L-Carnitine 4g

INTERVENTIONS:
Dietary Supplement: L-Carnitine 4g — 500ml enteral nutrition solution containing 4g of L-carnitine
  Arms: Enteral Nutrition with L-Carnitine
Dietary Supplement: Enteral Nutrition — Enteral nutrition was given 500 ml per day for a total of 84 days.
  Arms: Enteral nutrition

SUMMARY:
This is a multicenter, double-blind randomized controlled clinical study designed to evaluate the efficacy and safety of oral nutritional supplements (ONS) containing levocarnitine for cachexia in lung cancer patients scheduled for or undergoing chemotherapy.

Study Design:

Recruitment: Approximately 126 pathologically confirmed patients meeting the inclusion criteria will be enrolled across four hospitals (Army Characteristic Medical Center, Chongqing Fifth People's Hospital, Chongqing Thirteenth People's Hospital, and Chongqing Qianjiang District Central Hospital). The planned enrollment is 60 patients at Army Characteristic Medical Center, 22 at Chongqing Fifth People's Hospital, 22 at Chongqing Thirteenth People's Hospital, and 22 at Chongqing Qianjiang District Central Hospital.

Randomization: Patients will be randomly assigned in a 1:1 ratio to the control group (63 patients) or the intervention group (63 patients).

Interventions:

Control Group: Receive 500 mL of enteral nutrition solution daily for 12 weeks (84 days).

Intervention Group: Receive 500 mL of enteral nutrition solution containing 4 g of levocarnitine daily for 12 weeks (84 days).

Evaluations:

Efficacy Assessments: Body composition analysis and other evaluations will be conducted at baseline and after ONS treatment with levocarnitine to assess the effectiveness of the intervention.

Safety Assessments: Safety events during the levocarnitine-containing ONS treatment period and within 28 days after neoadjuvant therapy will be collected to evaluate treatment safety.

Follow-up: After chemotherapy, the investigator will determine the optimal adjuvant treatment and follow-up protocols to assess recurrence and survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 1. Primary lung tumor confirmed by cytology or histology; 2.Meeting the diagnostic criteria for cachexia (with one of the following criteria):

  1. Weight loss >5% in the past 6 months (without active weight loss);
  2. Body mass index (BMI) <20 and weight loss >2%;
  3. Decreased total skeletal muscle index (detected by bioelectrical impedance analysis: <7.26 kg/m² for males; <5.45 kg/m² for females) and weight loss >2%; 3.Age ≥18 years; 4.Patients scheduled to receive or currently undergoing chemotherapy; 5.Patients with an expected survival period ≥3 months; 6.Signed written informed consent and able to comply with the study visit schedule and relevant procedures; 7.Sufficient organ function before the first study treatment (no use of any blood components, leukocyte-elevating drugs, or platelet-elevating drugs within 14 days prior to randomization):

  <!-- -->

  1. Absolute neutrophil count ≥1.5×10⁹/L;
  2. Platelet count ≥100×10⁹/L;
  3. Hemoglobin >90 g/L;
  4. Serum creatinine <1.5×upper limit of normal (ULN) or creatinine clearance (CLcr) calculated by the Cockcroft-Gault formula >50 mL/min;
  5. Total bilirubin <1.5×ULN (for Gilbert syndrome patients, <3×ULN is acceptable);
  6. AST and ALT <2.5×ULN (for patients with liver metastases, ≤5×ULN);
  7. International normalized ratio (INR) or activated partial thromboplastin time (APTT) ≤1.5×ULN, unless the subject is receiving anticoagulant therapy

Exclusion Criteria:

* 1.Patients scheduled for lung cancer surgery within the next 3 months; 2.Patients with uncontrolled hyperglycemia after adequate treatment; 3.Patients allergic to levocarnitine; 4.Patients with contraindications to enteral nutrition, including but not limited to active gastrointestinal bleeding, complete intestinal obstruction, etc.; 5.Patients with diseases severely affecting digestion and absorption, including but not limited to subtotal gastrectomy, history of intestinal surgery, etc.; 6.Patients with clinically significant cardiovascular and cerebrovascular diseases, including but not limited to:

  1. Myocardial infarction or unstable angina within 6 months before the first drug administration;
  2. Stroke or transient ischemic attack within 6 months before the first drug administration;
  3. Hypertension that cannot be controlled after optimal antihypertensive treatment (systolic blood pressure >160 mmHg and/or diastolic blood pressure ≥100 mmHg);
  4. Patients with clinically significant arrhythmia who have been stable for >14 days before the first drug administration may be enrolled;
  5. Congestive heart failure (New York Heart Association [NYHA] functional classification > Class 3; see Appendix VI for details);
  6. Myocarditis; 7.Patients currently participating in interventional clinical research treatment, or who have received other investigational drugs or devices within 4 weeks prior to randomization; 8.Active tuberculosis or tuberculosis requiring medical intervention at the current stage, including but not limited to pulmonary tuberculosis; 9.Patients with known mental illnesses or substance abuse that may affect compliance with trial requirements, or a history of alcohol abuse; 10.Patients with medical history, diseases, treatments, or laboratory abnormalities that may interfere with trial results or prevent the subject from participating in the study throughout the process, or where the investigator deems participation not in the subject's best interest; 11.Local or systemic diseases caused by non-malignant tumors, or secondary reactions to cancer, which may lead to higher medical risks and/or uncertainty in survival evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Total Skeletal Muscle Mass | At enrollment, Day 21, Day 42, Day 63, Day 84, six months, and 12 months
  The total skeletal muscle mass (TSMM) is the primary endpoint of this study. It is defined as the total weight of skeletal muscles throughout the human body, typically expressed in kilograms (kg). This assessment is conducted using a body composition analyzer.

SECONDARY OUTCOMES:
BMI | At enrollment, Day 21, Day 42, Day 63, Day 84, six months, and 12 months
  The body mass index (BMI) is defined as a value obtained by dividing body weight (in kilograms) by the square of height (in meters). The formula is: weight / height²
Grip strength | At enrollment, Day 21, Day 42, Day 63, Day 84, six months, and 12 months
  It is defined as the force generated by the contraction of hand muscles. This force reflects the comprehensive strength level of hand flexor muscles (such as the flexor digitorum superficialis, flexor digitorum profundus, and flexor pollicis longus) and related muscle groups (such as the thenar muscles and hypothenar muscles). To some extent, it can reflect an individual's overall muscle strength and physical function status. This assessment is measured using an electronic grip dynamometer.
Inflammatory cytokines | At enrollment, Day 21, Day 42, Day 63, Day 84, six months, and 12 months
  Inflammatory molecules refer to a class of bioactive substances produced and released during the inflammatory response, which play a key role in the initiation, development, and regulation of inflammation. This assessment uses interleukin-1 (IL-1), interleukin-6 (IL-6), tumor necrosis factor-α (TNF-α), and C-reactive protein (CRP).
Nutritional Score | At enrollment, Day 21, Day 42, Day 63, Day 84, six months, and 12 months
  The nutritional score is defined as a quantitative method used to assess the nutritional status of individuals or groups, and this assessment is measured using PG-SGA and NRS2002.
Quality of Life Score | At enrollment, Day 21, Day 42, Day 63, Day 84, six months, and 12 months
  The quality of life score is a quantitative evaluation of the quality of life of individuals or groups, and this assessment is conducted using the EORTC QLQ-C30 C3.0 Chinese version (Quality of Life Questionnaire for Lung Cancer Patients).

CONTACTS AND LOCATIONS:
Overall Officials: hongxia Xu, Study Director — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Daping Hospital and the Research Institute of Surgery of The Third Military Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: Undecided